CLINICAL TRIAL: NCT05108194
Title: Feasibility of a Personalized Short Message Service Intervention for Insomnia
Brief Title: Feasibility of a Personalized SMS Intervention for Insomnia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Missouri, St. Louis (Other)
Responsible Party: Principal Investigator, Chelsey Wilks, Assistant Professor, University of Missouri, St. Louis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMissouriSL
Record Dates: First submitted 2021-10-11; First posted 2021-11-04 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Insomnia; Sleep Disorder
Keywords: Insomnia; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: All participants will enroll in the intervention after a two week assessment phase.
Masking Description: All participants will be enrolled in the intervention and all participants and study staff will be aware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1: Intervention (Experimental): Participants (N=50) who endorse insomnia will be followed for 8 weeks. All participants will be asked to download a separate app to passively monitor sleep that will inform the personalized messages. Participants will also be asked to respond to daily prompts in order to validate the passive sleep data. The study includes two phases: (1) a training and validation phase and (2) an intervention phase. During phase 1, participants' sleep habits and other behaviors will be monitored for two weeks in order to validate and optimize the SMS personalized sleep intervention (PSI). In phase 2, participants will be transitioned to the intervention phase of the study.
  Interventions: Behavioral: SMS Personalized Sleep Intervention

INTERVENTIONS:
Behavioral: SMS Personalized Sleep Intervention — All participants will be enrolled in the intervention to evaluate the feasibility and acceptability of the SMS-PSI. After the data training and validation phase, participants will be provided with at least one and up to three daily text messages that offer users a specific strategy based on strategies from CBTi. All participants will have access to a "user dashboard", which is a web-app that includes personalized sleep-tracking information and the opportunity to customize their messaging. The person-level acceptability and adherence to the sleep strategies will be evaluated via self-report endorsement from daily diary and whether users added suggestions to their calendars. Both adherence and acceptability will be collected and integrated with the selection algorithm to optimize subsequent SMS suggestions.

SUMMARY:
The goal of this research is to establish a proof of concept for optimizing and evaluating a personalized SMS intervention based for individuals with chronic sleep problems.

DETAILED DESCRIPTION:
Insomnia is a pervasive disorder affecting approximately 10-40% of the U.S. population in a given year. In addition, insomnia has been identified as a transdiagnostic symptom that cuts across numerous other psychological disorders. Interventions that target disordered sleep may attenuate symptomatic distress for a multitude of psychological disorders, making it a potentially potent intervention target with broad public health potential. Despite the ubiquity of the problem, only a fraction of individuals who could benefit actually receive the most effective intervention for insomnia, cognitive behavioral therapy for insomnia (CBT-I). Emerging research has pointed to the possibility of monitoring behavior and delivering personalized interventions to specific individuals via mobile devices. Personalized and adaptive interventions delivered via Short Message Service (SMS) provide a relatively simple solution to prompt individuals to engage in personalized interventions outside the context of opening or downloading a mobile mental health app. The content of text messages have the capacity to modulate behavior via prompts, motivational messages, and "nudges." By using brief, motivational messages based on evidence-based treatment for sleep (e.g. CBT-I), there is the potential to reduce dysfunctional sleep patterns at scale.

ELIGIBILITY:
Inclusion Criteria:

* clinical insomnia (defined by scoring ≥ 15 on the insomnia severity index)

Exclusion Criteria:

* under 18 y.o.
* unable to read or write in English
* do not own a Smart Phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | 8 weeks
  Insomnia severity

SECONDARY OUTCOMES:
System Usability Scale | 8 weeks
  Usability of the intervention

OTHER OUTCOMES:
PROMIS: Sleep related impairment | 8 weeks
  Sleep-related functional impairment
Flinders Fatigue Scale | 8 weeks
  Fatigue
Patient Health questionnaire 8 item | 8 weeks
  Depression
Difficulties in Emotion Regulation Scale | 8 weeks
  Emotion regulation

CONTACTS AND LOCATIONS:
Overall Officials: Chelsey R Wilks, PhD, Principal Investigator — University of Missouri, St. Louis
Locations (1):
- University of Missouri-St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant outcome data will be made available to other researchers upon approval of home institution ethics approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after data collection is complete
Access Criteria: Approval from home institution internal review board

REFERENCES:
- [Background] Mai E, Buysse DJ. Insomnia: Prevalence, Impact, Pathogenesis, Differential Diagnosis, and Evaluation. Sleep Med Clin. 2008;3(2):167-174. doi: 10.1016/j.jsmc.2008.02.001. No abstract available. PMID 19122760
- [Background] Dolsen EA, Asarnow LD, Harvey AG. Insomnia as a transdiagnostic process in psychiatric disorders. Curr Psychiatry Rep. 2014 Sep;16(9):471. doi: 10.1007/s11920-014-0471-y. PMID 25030972
- [Background] Britton PC, McKinney JM, Bishop TM, Pigeon WR, Hirsch JK. Insomnia and risk for suicidal behavior: A test of a mechanistic transdiagnostic model in veterans. J Affect Disord. 2019 Feb 15;245:412-418. doi: 10.1016/j.jad.2018.11.044. Epub 2018 Nov 5. PMID 30423469
- [Background] Cai GH, Theorell-Haglow J, Janson C, Svartengren M, Elmstahl S, Lind L, Lindberg E. Insomnia symptoms and sleep duration and their combined effects in relation to associations with obesity and central obesity. Sleep Med. 2018 Jun;46:81-87. doi: 10.1016/j.sleep.2018.03.009. Epub 2018 Apr 3. PMID 29773216
- [Background] Kyle SD, Morgan K, Espie CA. Insomnia and health-related quality of life. Sleep Med Rev. 2010 Feb;14(1):69-82. doi: 10.1016/j.smrv.2009.07.004. Epub 2009 Dec 4. PMID 19962922
- [Background] Morin CM, Rodrigue S, Ivers H. Role of stress, arousal, and coping skills in primary insomnia. Psychosom Med. 2003 Mar-Apr;65(2):259-67. doi: 10.1097/01.psy.0000030391.09558.a3. PMID 12651993
- [Background] Fortier-Brochu E, Beaulieu-Bonneau S, Ivers H, Morin CM. Insomnia and daytime cognitive performance: a meta-analysis. Sleep Med Rev. 2012 Feb;16(1):83-94. doi: 10.1016/j.smrv.2011.03.008. Epub 2011 Jun 1. PMID 21636297
- [Background] Margolies SO, Rybarczyk B, Vrana SR, Leszczyszyn DJ, Lynch J. Efficacy of a cognitive-behavioral treatment for insomnia and nightmares in Afghanistan and Iraq veterans with PTSD. J Clin Psychol. 2013 Oct;69(10):1026-42. doi: 10.1002/jclp.21970. Epub 2013 Apr 29. PMID 23629959
- [Background] Manber R, Edinger JD, Gress JL, San Pedro-Salcedo MG, Kuo TF, Kalista T. Cognitive behavioral therapy for insomnia enhances depression outcome in patients with comorbid major depressive disorder and insomnia. Sleep. 2008 Apr;31(4):489-95. doi: 10.1093/sleep/31.4.489. PMID 18457236
- [Background] Waite F, Myers E, Harvey AG, Espie CA, Startup H, Sheaves B, Freeman D. Treating Sleep Problems in Patients with Schizophrenia. Behav Cogn Psychother. 2016 May;44(3):273-87. doi: 10.1017/S1352465815000430. Epub 2015 Jul 30. PMID 26751571
- [Background] Trauer JM, Qian MY, Doyle JS, Rajaratnam SM, Cunnington D. Cognitive Behavioral Therapy for Chronic Insomnia: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Aug 4;163(3):191-204. doi: 10.7326/M14-2841. PMID 26054060
- [Background] Mitchell MD, Gehrman P, Perlis M, Umscheid CA. Comparative effectiveness of cognitive behavioral therapy for insomnia: a systematic review. BMC Fam Pract. 2012 May 25;13:40. doi: 10.1186/1471-2296-13-40. PMID 22631616
- [Background] Stinson K, Tang NK, Harvey AG. Barriers to treatment seeking in primary insomnia in the United Kingdom: a cross-sectional perspective. Sleep. 2006 Dec;29(12):1643-6. doi: 10.1093/sleep/29.12.1643. PMID 17252896
- [Background] Lattie EG, Schueller SM, Sargent E, Stiles-Shields C, Tomasino KN, Corden ME, Begale M, Karr CJ, Mohr DC. Uptake and Usage of IntelliCare: A Publicly Available Suite of Mental Health and Well-Being Apps. Internet Interv. 2016 May;4(2):152-158. doi: 10.1016/j.invent.2016.06.003. Epub 2016 Jun 16. PMID 27398319
- [Background] Lau PW, Lau EY, Wong del P, Ransdell L. A systematic review of information and communication technology-based interventions for promoting physical activity behavior change in children and adolescents. J Med Internet Res. 2011 Jul 13;13(3):e48. doi: 10.2196/jmir.1533. PMID 21749967
- [Background] Szaszi B, Palinkas A, Palfi B, Szollosi A, Aczel B. A Systematic Scoping Review of the Choice Architecture Movement: Toward Understanding When and Why Nudges Work: Systematic Scoping Review of the Nudge Movement. J Behav Decis Mak. 2018;31(3):355-366. http://doi:10.1002/bdm.2035
- [Background] Hardeman W, Houghton J, Lane K, Jones A, Naughton F. A systematic review of just-in-time adaptive interventions (JITAIs) to promote physical activity. Int J Behav Nutr Phys Act. 2019 Apr 3;16(1):31. doi: 10.1186/s12966-019-0792-7. PMID 30943983
- [Background] Hebert ET, Ra CK, Alexander AC, Helt A, Moisiuc R, Kendzor DE, Vidrine DJ, Funk-Lawler RK, Businelle MS. A Mobile Just-in-Time Adaptive Intervention for Smoking Cessation: Pilot Randomized Controlled Trial. J Med Internet Res. 2020 Mar 9;22(3):e16907. doi: 10.2196/16907. PMID 32149716
- [Background] Saeb S, Cybulski TR, Schueller SM, Kording KP, Mohr DC. Authorship Correction: Scalable Passive Sleep Monitoring Using Mobile Phones: Opportunities and Obstacles. J Med Internet Res. 2017 Apr 28;19(4):e143. doi: 10.2196/jmir.7932. PMID 30578218
- [Background] Wilks CR, Lungu A, Ang SY, Matsumiya B, Yin Q, Linehan MM. A randomized controlled trial of an Internet delivered dialectical behavior therapy skills training for suicidal and heavy episodic drinkers. J Affect Disord. 2018 May;232:219-228. doi: 10.1016/j.jad.2018.02.053. Epub 2018 Feb 17. PMID 29499504
- [Background] Schroeder J, Suh J, Wilks C, Czerwinski M, Munson SA, Fogarty J, Althoff T. Data-Driven Implications for Translating Evidence-Based Psychotherapies into Technology-Delivered Interventions. Int Conf Pervasive Comput Technol Healthc. 2020 May;2020:274-287. doi: 10.1145/3421937.3421975. PMID 33912357
- [Background] Wilks CR, Yin Q, Zuromski KL. User Experience Affects Dropout from Internet-Delivered Dialectical Behavior Therapy. Telemed J E Health. 2020 Jun;26(6):794-797. doi: 10.1089/tmj.2019.0124. Epub 2019 Sep 6. PMID 31502945
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Gradisar M, Lack L, Richards H, Harris J, Gallasch J, Boundy M, Johnston A. The Flinders Fatigue Scale: preliminary psychometric properties and clinical sensitivity of a new scale for measuring daytime fatigue associated with insomnia. J Clin Sleep Med. 2007 Dec 15;3(7):722-8. PMID 18198807
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Gratz KL, Roemer L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. J Psychopathol Behav Assess. 2004;26(1):41-54. http://doi:10.1023/B:JOBA.0000007455.08539.94
- [Background] Bangor A, Kortum PT, Miller JT. An Empirical Evaluation of the System Usability Scale. Int J Hum-Comput Interact. 2008;24(6):574-594. http://doi:10.1080/10447310802205776
- [Background] Mcmurtry SL, Hudson WW. The Client Satisfaction Inventory: Results of an Initial Validation Study. Res Soc Work Pract. 2000;10(5):644-663. http://doi:10.1177/104973150001000506
- [Background] Horvath AO, Greenberg LS. Development and validation of the Working Alliance Inventory. J Couns Psychol. 1989;36(2):223-233. http://doi:10.1037/0022-0167.36.2.223